CLINICAL TRIAL: NCT05207605
Title: Effects of Rhythmic Stabilization and Mckenzie Techniques on Pain and Function in Patients With Non-specific Chronic Low Back Pain
Brief Title: Effects of Rhythmic Stabilization and Mckenzie Techniques on Non Specific Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/21/0121
Record Dates: First submitted 2022-01-24; First posted 2022-01-26 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Back Pain
Keywords: non specific low back pain; paraspinal muscles
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhythmic Stabilization (RS) (Experimental): The patient is in sitting position and faces the physical therapist. The RST program consisted of alternating (trunk flexion-extension) isometric contractions against resistance for 10 seconds, with no motion intended
  Interventions: Other: Rhythmic Stabilization (RS)
- McKenzie technique (Experimental): McKenzie exercises will be guided to conduct four extension exercises and three flexion exercises.
  Interventions: Other: McKenzie technique

INTERVENTIONS:
Other: Rhythmic Stabilization (RS) — Group A includes rhythmic stabilization technique. The patient is in sitting position and faces the physical therapist. The RST program consisted of alternating (trunk flexion-extension) isometric contractions against resistance for 10 seconds, with no motion intended. Subjects performed 3 sets of 15 repetitions at maximal resistance provided by the same physical therapist. Rest intervals of 30 seconds and 60 seconds were provided after the completion of 15 repetitions for each pattern and between sets, respectively. The total duration of RS will be of approximately 33 minutes
  Arms: Rhythmic Stabilization (RS)
Other: McKenzie technique — McKenzie technique will be guided to conduct four extension exercises and three flexion exercisesAll flexion exercises will be repeated for ten repetitions for two sets. There are three minutes for resting intervals in every set. The McKenzie treatment will lasted for 20-40 minutes.
  Arms: McKenzie technique

SUMMARY:
Non-speciﬁc low back pain is deﬁned as low back pain not attributable to an identifiable, known speciﬁc pathology. Non-specific low back pain accounts for over 90% of patients presenting to primary care and these are the majority of the individuals with low back pain that present to physiotherapy.Objective of this study is to compare the effects of rhythmic stabilization and McKenzie technique on pain and function in patients with non-specific chronic low back pain

DETAILED DESCRIPTION:
Low back pain is the most common musculoskeletal condition worldwide. About 18% of the world's population suffers from low back pain and approximately 39% will suffer at least one episode of low back pain in their lifetime. Consequently, the costs associated with the treatment of patients with low back pain, absence from work , and disability are extremely high. The annual worldwide LBP incidence in adults to be 15% and the point prevalence to be 30% .A sedentary lifestyle with a lack of physical activity results in the loss of muscle power and strength and can be a predictor of LBP leading to recurrent LBP .In addition, a specific diagnosis of low back pain cannot be obtained in approximately 80% patients with low back pain, indicating that patients with low back pain are often diagnosed with nonspecific low back pain. Non-specific chronic low back pain (LBP) is a rather common and predominant health problem worldwide that affects people of all ages. Nonspecific low back pain is defined in the European guidelines for the management of chronic nonspecific low back pain (CNSLBP) as low back pain that is not attributable to a recognizable, specific pathology (e.g., infection, tumor, osteoporosis, fracture, structural deformity, and inflammatory diseases, such as ankylosing spondylitis, radicular syndrome, and cauda equina syndrome)Characteristic of chronic nonspecific low back pain are heavy pain, worsening with exertion and relieve with rest. In some cases the cause may be sprain or overstretch of a ligament or muscles. The endurance of trunk muscles is low in patients with low back pain as compared to individual without low back pain. The deep trunk muscles (Transverse Abdominis and Multifidus) responsible for maintaining the stability of spine. In other cases the cause may be a minor problem with the disc between two vertebrae or a minor problem with a small facet joint between two vertebrae. There may be other minor problems in the structures and tissues of the lower back that result in pain.The terminology becomes "chronic" low back pain when the symptom duration exceeds three months (nCLBP).Chronic low back pain (LBP) represents a significant healthcare problem that results in substantial costs to society .It is a prevalent condition that leads to increased disability and decreased quality of life.Non-specific LBP belongs to the group of musculoskeletal disorders, which include diverse conditions affecting muscles, bones, and/or joints of the limbs or the spine.

ELIGIBILITY:
Inclusion Criteria:

* NSCLBP patients aged ≥ 18 to 45 years old(23).
* Both genders.
* Mild to moderate back pain with NPRS pain score value of between 2/10 - 6/10.
* Pain from at least past three months (12 weeks).
* No radiating pain below the gluteal fold.

Exclusion Criteria:

* Diagnosis of systemic metabolic and/or neurological disorder.
* Neuropathic pain.
* Any referred pain below gluteal fold or neurological involvement in lower limbs is not included.
* Pathological conditions or diagnosed with disk herniation, spinal stenosis, spondylolysthesis, and spondylitis and other medical illnesses such as tumor, kidney disease, and visceral disease that can be related with low back pain excluded in this study.
* Participants who had undergone surgery for LBP.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-06-12 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NPRS) | 4th week
  Numeric Rating Scale (NPRS) is most frequently used instruments to measure pain intensity in low back pain (LBP).The 11-point numeric with 0 representing No pain, 1-3 representing Mild Pain (nagging, annoying, interfering little with ADLs), 4-6 representing Moderate Pains (interferes significantly with ADLs), 7-10 representing Sever Pain (disabling, unable to perform ADLs)
Oswestery Disability Index | 4th week
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools. This scale contain question related to functional activities of pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and travelling. For patients understanding, URDU version is used. Interpretation of scale are 0% to 20% for minimal disability, 21% to 40% for moderate disability, 41 % to 60 % for severe disability 61% to 80 % for crippled and 81 % to 100 %. Bed-bound

SECONDARY OUTCOMES:
ROM lumber spine (flexion) | 4th week
  The spinous process of the 1st sacral vertebra and the 12th thoracic vertebra will be considered as reference points for measuring the range of motion in bending forward
ROM lumber spine (extension) | 4th week
  The spinous process of the 1st sacral vertebra and the 12th thoracic vertebra will be considered as reference points for measuring the range of motion in bending backward
ROM lumber spine (side flexion) | 4th week
  The spinous process of the 12th thoracic vertebra was considered as reference point for measuring the range of motion of lumbar side flexion

CONTACTS AND LOCATIONS:
Overall Officials: Sana Hafeez, PhD*, Principal Investigator — Riphah International University Lahore Campus
Locations (1):
- Riphah international university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luz Junior MAD, Almeida MO, Santos RS, Civile VT, Costa LOP. Effectiveness of Kinesio Taping in Patients With Chronic Nonspecific Low Back Pain: A Systematic Review With Meta-analysis. Spine (Phila Pa 1976). 2019 Jan 1;44(1):68-78. doi: 10.1097/BRS.0000000000002756. PMID 29952880
- [Background] Ganesan S, Acharya AS, Chauhan R, Acharya S. Prevalence and Risk Factors for Low Back Pain in 1,355 Young Adults: A Cross-Sectional Study. Asian Spine J. 2017 Aug;11(4):610-617. doi: 10.4184/asj.2017.11.4.610. Epub 2017 Aug 7. PMID 28874980
- [Background] Citko A, Gorski S, Marcinowicz L, Gorska A. Sedentary Lifestyle and Nonspecific Low Back Pain in Medical Personnel in North-East Poland. Biomed Res Int. 2018 Sep 9;2018:1965807. doi: 10.1155/2018/1965807. eCollection 2018. PMID 30271778
- [Background] Yang JH, Suk KS, Lee BH, Jung WC, Kang YM, Kim JH, Kim HS, Lee HM, Moon SH. Efficacy and Safety of Different Aceclofenac Treatments for Chronic Lower Back Pain: Prospective, Randomized, Single Center, Open-Label Clinical Trials. Yonsei Med J. 2017 May;58(3):637-643. doi: 10.3349/ymj.2017.58.3.637. PMID 28332372
- [Background] Iizuka Y, Iizuka H, Mieda T, Tsunoda D, Sasaki T, Tajika T, Yamamoto A, Takagishi K. Prevalence of Chronic Nonspecific Low Back Pain and Its Associated Factors among Middle-Aged and Elderly People: An Analysis Based on Data from a Musculoskeletal Examination in Japan. Asian Spine J. 2017 Dec;11(6):989-997. doi: 10.4184/asj.2017.11.6.989. Epub 2017 Dec 7. PMID 29279756
- [Background] Imamura M, Alfieri FM, Filippo TR, Battistella LR. Pressure pain thresholds in patients with chronic nonspecific low back pain. J Back Musculoskelet Rehabil. 2016 Apr 27;29(2):327-336. doi: 10.3233/BMR-150636. PMID 26406214